CLINICAL TRIAL: NCT00356356
Title: Open-label, Long-term Extension Study of Etanercept in the Treatment of Patients With Ankylosing Spondylitis Who Participated in Protocol 16.0037
Brief Title: 16.0040 Ankylosing Spondylitis Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20021640; 016.0040
Record Dates: First submitted 2006-07-24; First posted 2006-07-26 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

ARMS (1):
- All subjects (Experimental): 257 subjects
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Etanercept 50 mg/wk administered as 2-25 mg SQ injections at separate injection sites

SUMMARY:
The purpose of this study was to evaluate extended safety and efficacy of etanercept in adults with Ankylosing Spondylitis.

DETAILED DESCRIPTION:
This multicenter, open-label extension study will evaluate the safety and clinical benefit of etanercept in the treatment of Ankylosing Spondylitis in subjects previously enrolled in Protocol 16.0037.

ELIGIBILITY:
Inclusion Criteria: - Subjects completing 24 weeks of study drug in protocol 16.0037 qualify to enroll into this study Other patients to meet the following criteria:

* Negative pregnancy test
* Subjects agree to use appropriate contraception throughout study
* Should be able to self-inject study drug or have someone who can do so
* Capable of understanding protocol and willing to provide written informed consent

Exclusion Criteria:

* Any change in NSAID or prednisone dose within 2 weeks of baseline
* Any change in hydroxychloroquine, sulfasalazine, or MTX dose within 4 weeks of baseline
* Use of DMARDs other than those mentioned above, within 4 weeks of enrollment
* Previous receipt of ani-TNF agents, other than etanercept
* Receipt of any other investigational drug within 30 days of baseline
* Grade 3 or 4 adverse event attributed to etanercept which recurred when etanercept was resumed
* Abnormality in chemistry or hematology profiles or significant concurrent medical events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2002-04; Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Treatment Response (using ASAS criteria) of at least 20% and absolute improvement of at least 10 units on a 0-100 scale in at least 3 of the 4 domains | Up to 4 years
Absence of deterioration (using ASAS criteria) of at least 20% and absolute improvement of at least 10 units on a 0-100 scale in the potential remaining ASAS domain | Up to 4 years

SECONDARY OUTCOMES:
DXA and MRI scans (at selected sites) | Up to 144 weeks
X-rays of cervical spine and lumbosacral spine | Up to 4 years
Type and grade of toxicities | Up to 4 years
ASAS Response Criteria at weeks 24, 36, 48, 60, 72, 84, 96, 108, 120, and the ASAS Response Criteria at 50% and 70% levels at weeks 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, and 144. | Up to 4 years
Frequency and time to partial remission as defined in Anderson, 2001: Value of <20 (on a scale of 0-100) in each of the following 4 domains: VAS Patient Global Assessment, VAS Pain Score, BASFI, and BASDAI morning stiffness-related scores | Up to 4 years
Spinal mobility measured with Schober's test, chest expansion, and occiput to wall distance | Up to 120 weeks
Complete joint assessment | Up to 120 weeks
Laboratory assessment of inflammation using CRP | Up to 120 weeks
Ability to reduce and discontinue concomitant NSAIDs, prednisone, hydroxychloroquine, sulfasalazine, and methotrexate | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Baraliakos X, Brandt J, Listing J, Haibel H, Sorensen H, Rudwaleit M, Sieper J, Braun J. Outcome of patients with active ankylosing spondylitis after two years of therapy with etanercept: clinical and magnetic resonance imaging data. Arthritis Rheum. 2005 Dec 15;53(6):856-63. doi: 10.1002/art.21588. PMID 16342093
- [Result] Boonen A, Patel V, Traina S, Chiou CF, Maetzel A, Tsuji W. Rapid and sustained improvement in health-related quality of life and utility for 72 weeks in patients with ankylosing spondylitis receiving etanercept. J Rheumatol. 2008 Apr;35(4):662-7. Epub 2008 Feb 15. PMID 18278836
- [Result] Davis JC, van der Heijde DM, Braun J, Dougados M, Cush J, Clegg D, Inman RD, Kivitz A, Zhou L, Solinger A, Tsuji W. Sustained durability and tolerability of etanercept in ankylosing spondylitis for 96 weeks. Ann Rheum Dis. 2005 Nov;64(11):1557-62. doi: 10.1136/ard.2004.035105. Epub 2005 Apr 20. PMID 15843448
- [Result] Davis JC Jr, van der Heijde DM, Braun J, Dougados M, Clegg DO, Kivitz AJ, Fleischmann RM, Inman RD, Ni L, Lin SL, Tsuji WH. Efficacy and safety of up to 192 weeks of etanercept therapy in patients with ankylosing spondylitis. Ann Rheum Dis. 2008 Mar;67(3):346-52. doi: 10.1136/ard.2007.078139. Epub 2007 Oct 29. PMID 17967833
- [Derived] Baraliakos X, Szumski AE, Kwok KK, Vlahos B, Borlenghi CE. Long-term Etanercept Response for Patients with Radiographic Axial Spondyloarthritis Based on Achievement of Early, Intermediate, or Late Responses During Index Studies. Rheumatol Ther. 2024 Jun;11(3):583-597. doi: 10.1007/s40744-024-00656-3. Epub 2024 Mar 15. PMID 38488976
- [Derived] Baraliakos X, Szumski A, Koenig AS, Jones H. The role of C-reactive protein as a predictor of treatment response in patients with ankylosing spondylitis. Semin Arthritis Rheum. 2019 Jun;48(6):997-1004. doi: 10.1016/j.semarthrit.2018.10.019. Epub 2018 Nov 2. PMID 30473179
- [Derived] van der Heijde D, Landewe R, Einstein S, Ory P, Vosse D, Ni L, Lin SL, Tsuji W, Davis JC Jr. Radiographic progression of ankylosing spondylitis after up to two years of treatment with etanercept. Arthritis Rheum. 2008 May;58(5):1324-31. doi: 10.1002/art.23471. PMID 18438853
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/